CLINICAL TRIAL: NCT05707871
Title: Cardiovascular Effects of Very Low Nicotine Content Cigarettes
Acronym: CEV
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00092813
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Use
Keywords: Cigarette smoking; Nicotine Content; Cardiovascular Disorders
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Within Subject
Who Masked: Participant
Masking Description: Participants will be blinded to content of nicotine in cigarettes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Brand of Cigarettes (Active Comparator): Participants will smoke 2-3 cigarettes of their usual brand
  Interventions: Other: usual brand of Cigarettes
- Research Cigarettes (SPECTRUM) (Experimental): Participants will smoke 1-2 SPECTRUM cigarettes
  Interventions: Drug: SPECTRUM cigarettes

INTERVENTIONS:
Drug: SPECTRUM cigarettes — SPECTRUM cigarettes have varying amount of nicotine content
  Other Names: Cigarette Smoke
  Arms: Research Cigarettes (SPECTRUM)
Other: usual brand of Cigarettes — Usual Brand of Cigarettes
  Arms: Usual Brand of Cigarettes

SUMMARY:
The study is measuring Cardiovascular effects of very low nicotine content cigarettes on daily and non-daily smokers

DETAILED DESCRIPTION:
The FDA is planning regulatory actions to limit nicotine levels in cigarettes as far as it is not reduced to zero. The strategy is designed to reduce the addictiveness of cigarettes. However, nicotine related effects of the cigarettes with reduced nicotine content on various body systems are largely unknown. Following formal implementation of the regulatory policy what cardiovascular effects of reduced nicotine cigarettes, also called very low nicotine content cigarettes (VLNCC) are expected to persist is important to determine. This study will determine the cardiovascular effects of VLNCC such as change in heart rate, autonomic functions and indices of ventricular repolarization in smokers. Participants will be asked to smoke two VLNCC and one normal nicotine content cigarette (NNCC) while we will be recording their electrocardiogram (ECG) to see a change in heart rate, heart rate variability and indices of ventricular repolarization.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported cigarette smoking at least once in the past 30 days
* ≥21 years old
* Willingness to smoke research cigarettes or usual brand cigarettes during lab visit.
* Ability to speak, comprehend, and read English sufficiently to complete study procedures

Exclusion Criteria:

* Self-reported diagnosis of cardiovascular diseases like coronary artery disease, stroke, peripheral artery disease, cardiac arrhythmia, pulmonary embolism & blood clots in legs and arm in the past 3 months
* Body temperature ≥ 100.4˙F
* Unstable health conditions interfering with electrocardiogram (ECG) measurements
* Self-reported diagnosis of hyperthyroidism or thyrotoxicosis
* Currently pregnant (as indicated by urine pregnancy test at the start of laboratory visit) or breastfeeding.
* Currently seeking treatment to quit smoking

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Heart rate - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC102/103(0.5mg nicotine) | Hour 1
  Change in heart rate from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC)s - NRC102/103(0.5mg nicotine)
Change in Heart rate - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC301/302(2.4mg nicotine) | Hour 1
  Change in heart rate from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC)s - NRC301/302(2.4mg nicotine)
Change in Heart rate - Normal Nicotine Content Cigarettes (NNCC)s - NRC600/601(15.8mg nicotine) | Hour 1
  Change in heart rate from pre-exposure to post-exposure for the normal nicotine content cigarettes (NNCC)s - NRC600/601(15.8mg nicotine)

SECONDARY OUTCOMES:
Change in Heart rate variability(HRV) - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC102/103(0.5mg nicotine) | Hour 1
  Change in measures of heart rate variability (HF, LF, LF/HF, RMSSD = root mean square of standard deviation; SDNN = standard deviation of normal-to-normal intervals, Total power) from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC)s
Change in Heart rate variability(HRV) - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC301/302(2.4mg nicotine) | Hour 1
  Change in measures of heart rate variability (HF, LF, LF/HF, RMSSD = root mean square of standard deviation; SDNN = standard deviation of normal-to-normal intervals, Total power) from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC)s
Change in Heart rate variability(HRV) - Normal Nicotine Content Cigarettes (NNCC)s - NRC600/601(15.8mg nicotine) | Hour 1
  Change in measures of heart rate variability (HF, LF, LF/HF, RMSSD = root mean square of standard deviation; SDNN = standard deviation of normal-to-normal intervals, Total power) from pre-exposure to post-exposure for the Normal Nicotine Content Cigarettes (NNCC)s
Change in electrocardiogram (ECG) Measures - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC102/103(0.5mg nicotine) | Hour 1
  Measures of ventricular repolarization (Q-T interval, QTc, Tp-e interval)from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC)s
Change in electrocardiogram (ECG) Measures - Very Low Nicotine Content Cigarettes (VLNCC)s - NRC300/301(2.4mg nicotine) | Hour 1
  Measures of ventricular repolarization (Q-T interval, QTc, Tp-e interval)from pre-exposure to post-exposure for the Very Low Nicotine Content Cigarettes (VLNCC) s
Change in electrocardiogram (ECG) Measures - Normal Nicotine Content Cigarettes (NNCC)s - NRC600/601(15.8mg nicotine) | Hour 1
  Measures of ventricular repolarization (Q-T interval, QTc, Tp-e interval)from pre-exposure to post-exposure for the Normal Nicotine Content Cigarettes (NNCC)s

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Donny, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benowitz NL, Henningfield JE. Establishing a nicotine threshold for addiction. The implications for tobacco regulation. N Engl J Med. 1994 Jul 14;331(2):123-5. doi: 10.1056/NEJM199407143310212. No abstract available. PMID 7818638
- [Background] Benowitz NL, Henningfield JE. Reducing the nicotine content to make cigarettes less addictive. Tob Control. 2013 May;22 Suppl 1(Suppl 1):i14-7. doi: 10.1136/tobaccocontrol-2012-050860. PMID 23591498
- [Background] Hatsukami DK, Kotlyar M, Hertsgaard LA, Zhang Y, Carmella SG, Jensen JA, Allen SS, Shields PG, Murphy SE, Stepanov I, Hecht SS. Reduced nicotine content cigarettes: effects on toxicant exposure, dependence and cessation. Addiction. 2010 Feb;105(2):343-55. doi: 10.1111/j.1360-0443.2009.02780.x. PMID 20078491
- [Background] Tachmes L, Fernandez RJ, Sackner MA. Hemodynamic effects of smoking cigarettes of high and low nicotine content. Chest. 1978 Sep;74(3):243-6. doi: 10.1378/chest.74.3.243. PMID 688779
- [Background] Moheimani RS, Bhetraratana M, Peters KM, Yang BK, Yin F, Gornbein J, Araujo JA, Middlekauff HR. Sympathomimetic Effects of Acute E-Cigarette Use: Role of Nicotine and Non-Nicotine Constituents. J Am Heart Assoc. 2017 Sep 20;6(9):e006579. doi: 10.1161/JAHA.117.006579. PMID 28931527